CLINICAL TRIAL: NCT06494072
Title: Short Versus Standard of Care Antibiotic Duration for Hospitalized Children With Uncomplicated Community-acquired Pneumonia: a Non-inferiority, Randomized Controlled Trial.
Brief Title: Short Versus Standard of Care Antibiotic Duration for Children Hospitalized for CAP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michelle Mitchell, Associate Professor of Pediatric Infectious Diseases, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00046965
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Community Acquired Pneumonia in Children
Keywords: inpatient; pediatric; hospitalized; community acquired pneumonia.; antibiotic duration
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Ampicillin; Injections; Ceftriaxone; Amoxicillin; sultamicillin; Amoxicillin-Potassium Clavulanate Combination; Clindamycin; Cefprozil; Levofloxacin

STUDY DESIGN:
Intervention Model Description: Comparison of short duration (5 days) versus a standard of care duration of antibiotics on the effective treatment of children hospitalized for uncomplicated community acquired pneumonia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short course antibiotic duration (Experimental): The participants in this group will receive a total antibiotic course of 5 days including the number of days received during their hospital admission and following hospital admission combined.
  Interventions: Drug: Ampicillin for Injection; Drug: Ceftriaxone for Injection; Drug: Amoxicillin; Drug: Ampicillin / Sulbactam Injection; Drug: Amoxicillin-clavulanate; Drug: Clindamycin; Drug: Cefprozil; Drug: Levofloxacin
- Standard of care antibiotic duration (Active Comparator): Participants will receive the standard-of-care antibiotic course in this group. That is, the duration of antibiotics will be decided by the primary treating physician in this group. The antibiotic course will include the number of days received during the participant's hospital admission and following hospital admission combined.
  Interventions: Drug: Ampicillin for Injection; Drug: Ceftriaxone for Injection; Drug: Amoxicillin; Drug: Ampicillin / Sulbactam Injection; Drug: Amoxicillin-clavulanate; Drug: Clindamycin; Drug: Cefprozil; Drug: Levofloxacin

INTERVENTIONS:
Drug: Ampicillin for Injection — Ampicillin is an intravenous antibiotic commonly used in the initial treatment of children hospitalized with community-acquired pneumonia.
Drug: Ceftriaxone for Injection — Ceftriaxone is an intravenous antibiotic commonly used in the initial treatment of children hospitalized with community-acquired pneumonia.
  Other Names: Rocephin
Drug: Amoxicillin — Amoxicillin is an oral antibiotic commonly used in the treatment of children hospitalized with community-acquired pneumonia to complete the antibiotic course after discharge.
Drug: Ampicillin / Sulbactam Injection — Ampicillin/Sulbactam is an intravenous antibiotic commonly used in the initial treatment of children hospitalized with community-acquired pneumonia.
  Other Names: Unasyn
Drug: Amoxicillin-clavulanate — Amoxicillin-clavulanate is an oral antibiotic commonly used in the treatment of children hospitalized with community-acquired pneumonia to complete the antibiotic course after discharge.
  Other Names: Augmentin
Drug: Clindamycin — Clindamycin is an antibiotic that can be given intravenously or orally that is sometimes used in the treatment of children hospitalized or discharged with community-acquired pneumonia.
  Other Names: Cleocin
Drug: Cefprozil — Cefprozil is an oral antibiotic sometimes used in the treatment of children hospitalized with community-acquired pneumonia to complete the antibiotic course after discharge.
  Other Names: Cefzil
Drug: Levofloxacin — Levofloxacin is an antibiotic that can be given intravenously or orally that is sometimes used in the treatment of children hospitalized or discharged with community-acquired pneumonia.
  Other Names: Levaquin

SUMMARY:
The goal of this open label, randomized, non-inferiority clinical trial is to compare the treatment success of a 5 day antibiotic course versus a standard antibiotic course (usually 7-14 days of antibiotics) in hospitalized children aged 3 months to 18 years, with uncomplicated community acquired pneumonia.

The main questions it aims to answer are:

* Does a 5 day course work as well as standard (longer) courses of antibiotics for treating community acquired pneumonia in children?
* Does a 5 day course cause less antibiotic side effects compared to a standard (longer) course of antibiotics in children with community acquired pneumonia?

Participants will

* be randomly assigned to either receive 5 total days or a total duration decided by the treating physician
* receive a brief follow up questionnaire regarding clinical symptoms, follow up care/antibiotics, and side effects via phone or email at days 5 and 14 from the start of antibiotics

Researchers will compare the experimental group (receiving 5 days duration) with the control group (standard duration) to see if 5 days is as successful as a standard duration.

DETAILED DESCRIPTION:
This is an open label, randomized, non-inferiority clinical trial to determine if a 5-day antibiotic course works as well compared to a standard antibiotic course (usually 7-10 days of antibiotics) in hospitalized children who are aged 3 months to less than 18 years old, with uncomplicated community acquired pneumonia.

We will recruit 150 participants meeting inclusion/exclusion criteria. Participants will be randomized to one of the study groups. In the experimental group, the participant will receive a total antibiotic course of 5 days. In the other group (control group), participants will receive the standard-of-care antibiotic course (the duration will be decided by the primary treating physician in this group). The selection of antibiotic therapy will be made by the treating physician, generally in accordance with the institutional clinical practice guideline on community acquired pneumonia, prior to enrollment in the study. Other medical care, aside from the treatment duration, will be the same and will be guided by the primary treating doctor. The primary treating doctor will also decide when the participant is medically ready for discharge from the hospital.

During the consenting process, a member of the research team will verify the contact numbers or email of the parent(s)/guardian of participant to be used after discharge for follow-up communication. Every participant's parent/guardian will receive a text message/email questionnaire on day 5 and day 14 after the start of antibiotics to assess for clinical improvement, side effect(s) to the antibiotics, recurrence of fever, or need for additional antibiotics or other medical care. Participants parent(s)/guardian will be contacted by phone for additional information if there is concern for a failure or significant medical concern.

The primary objective of this study is to compare the failure rate between a short course (5-days) and standard antibiotic course (usually 7-10 days of antibiotics) of antibiotics in hospitalized children with uncomplicated pneumonia. Failure will be defined as the clinical need for additional antibiotic treatment, emergency department visit or readmission to the hospital for a suspected lower respiratory tract infection within 14 days of treatment initiation.

The secondary objective will compare the rate of adverse drug events between short and long-course durations of antibiotic therapy in children hospitalized for CAP. Adverse drug events include any allergic reaction such as skin rash, itching or other and/or abdominal symptoms such as vomiting, stomach pain and diarrhea.

Data will be summarized by n (%) or mean and standard deviation (SD) or median and interquartile range (IQR). Continuous variables will be compared by t-test while categorical variables will be compared by Chi-square or Fisher's exact test. A 95% CI will be calculated for the difference in failure rate between the shorter antibiotic course (5-day) group and the standard course group. Non-inferiority will be declared if the 95% CI lies below 10%. P<0.05 will be considered statistically significant. Data will be analyzed by SAS version 9.4 (SAS Institute Inc., Cary, NC) and SPSS version 28.0 (IBM Corp., Armonk, NY).

ELIGIBILITY:
Inclusion Criteria (ALL of the following must be met):

1. Children aged 3 months to <18 years old
2. Hospitalized in either the acute care or the pediatric intensive care units
3. Clinically diagnosed with uncomplicated bacterial community acquired pneumonia (as determined by the treating physician)
4. Radiological findings suggestive of pneumonia (such as consolidation, lobar or interstitial infiltrates)
5. Achieved clinical stability within 72 hours from the first antibiotic dose (clinical stability includes being off supplemental oxygen/ventilatory support and temperature remaining < 38 Celsius).

Exclusion Criteria (presence of ANY of the following will exclude a potential participant):

1. Hemodynamic instability at any point during hospitalization that required inotropic support
2. Requirement of respiratory support > 72 hours
3. Presence of a parapneumonic effusion >10 mm on decubitus x-ray or greater than ¼ of hemithorax opacified on chest imaging
4. Need for chest tube placement
5. Extrapulmonary involvement (ie: another infection located outside of the lungs) except for otitis media if the planned treatment is ≤ 5 days
6. Pneumonia caused by known staphylococcus aureus identified from culture (blood, bronchoalveolar aspirate, tracheal aspirate, or pleural fluid)
7. Antibiotic course started >72 hours after admission
8. Antibiotics used for > 24 hours within the 2 weeks prior to admission
9. Chronic respiratory illness other than asthma or reactive airway disease
10. Immunocompromised patient (primary or secondary)
11. Primary physician refusal
12. Parent refusal
13. Non-English speakers
14. Pregnant or lactating female
15. Participant will become ≥ 18 years old at or before the time of day 14 follow up
16. Inability to adhere to follow up

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate | 14 days from the first dose antibiotics
  Treatment failure is defined as the clinical need for additional antibiotic treatment, an emergency department (ED) visit, or readmission to the hospital for a suspected lower respiratory tract infection within 14 days of treatment initiation.

SECONDARY OUTCOMES:
Adverse drug event rate | 14 days from the first dose antibiotics
  Adverse drug events include allergic reactions, skin rash, abdominal symptoms (such as vomiting, stomach pain, or diarrhea), or other plausible associated complaints described by the parent(s)/guardian.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mitchell, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Childrens Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated data results will be provided.